CLINICAL TRIAL: NCT01550796
Title: Treatment of Chronic Bothersome Tinnitus Using Cognitive Training and D-cycloserine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Director of Clinical Outcomes Research Office, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201110105
Record Dates: First submitted 2012-01-25; First posted 2012-03-12 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Tinnitus
Keywords: Tinnitus; Brain Fitness Program; Posit Science; D-cycloserine; Cognitive Training
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- d-cycloserine (Active Comparator): d-cycloserine 250 mg two days per week one hour prior to(cognitive training)
  Interventions: Behavioral: Cognitive Training
- Placebo (Placebo Comparator): Placebo pill two days per week 1 hour prior to cognitive training
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — 250 mg d-cycloserine or placebo taken orally one hour before Brain Fitness Program
  Other Names: Posit Science, Brain Fitnesss Program

SUMMARY:
The purpose of this research study is to determine if a medication along with a computer program designed to improve memory and other mental processes can help people like yourself with tinnitus. The medication that will be investigated, d-cycloserine, was developed as an antibiotic. However, more recently, research in other studies has shown that this medication may enhance learning and memory. The investigators would like to determine if computer programs designed to improve memory and attention are enhanced by this medication. In addition, the investigators hope to learn if the use of these programs can help participants with their tinnitus as well as their ability to remember and focus. All research participants will receive therapy with a computer-based program designed to improve memory and attention. Half of participants will also receive d-cycloserine while the other half of participants will receive placebo. The placebo is a sugar pill without active medication.

DETAILED DESCRIPTION:
Tinnitus is the perception of a "ringing or hissing" sound in the absence of an acoustic stimulus affecting more than 40 million people in the United States. While the exact etiology of chronic bothersome tinnitus is unknown, current evidence based on numerous studies and neuroimaging results suggests chronic bothersome tinnitus involves the central nervous system with abnormalities in neural networks including attention and emotional networks. These neuroplastic changes in multiple neural networks may offer targets in the treatment of chronic bothersome tinnitus.

The Brain Fitness Program® (Posit Science Corporation, San Francisco, California) is a cognitive rehabilitation program that has been used in the treatment of schizophrenia and geriatric populations, and has been shown to have favorable results by reorganizing aberrant neural networks. Preliminary results from our team have shown improvements in tinnitus severity and cognitive functioning for participants with chronic bothersome tinnitus using this cognitive rehabilitation program.

Recent studies in numerous disorders have shown d-cycloserine (DCS) augments learning therapy programs by enhancing neuroplasticity. In addition, the adjuvant use of DCS with learning therapies has been found to accelerate symptom reduction decreasing the time-burden needed for learning therapies. Based on the belief that chronic bothersome tinnitus involves changes in malleable neural networks that can be targets of therapy and that DCS enhances neuroplasticity, the investigators hypothesize that adjuvant DCS with cognitive rehabilitation treatment may improve tinnitus severity and the cognitive deficits associated with chronic bothersome tinnitus.

This randomized-controlled trial will use an abbreviated cognitive rehabilitation program given for 5 weeks with DCS or placebo to evaluate the impact of a neuroplasticity-sensitizing drug on tinnitus symptom severity and cognitive performance among patients with chronic bothersome tinnitus. A positive result on this study will have numerous implications, including offering a new treatment option for chronic bothersome tinnitus with few known side effects and limited time commitment or cost.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 35 and 65.
* Participants must have subjective, unilateral or bilateral, non-pulsatile tinnitus for at least a duration of 6 consecutive months.
* Participants must have bothersome tinnitus as defined by a THI ≥ 30.
* Participants must have access to a computer for at least 60 minutes per day, 2 days per week, for five consecutive weeks.
* Participants must be willing to work on the Brain Fitness Program® that will be provided at least 60 minutes per day, 2 days per week, for 5 consecutive weeks.
* Participants must be willing to return for two treatment study visits during the first week after enrollment in the study and an additional study visit after 5 weeks.
* Participants must be willing to complete the Brain Fitness Program® and other assessments as prescribed.
* Participants must be able to read, write, and speak English fluently as the Brain Fitness Program, tinnitus assessments, and neurocognitive testing are written and administered in English.
* Women of child-bearing age must agree to use a study-approved form of contraception and agree to not try to become pregnant during the duration of the study. If a participant becomes pregnant, they should inform the PI and will be immediately withdrawn from the study.
* Participants must be able to provide valid informed consent.

Exclusion Criteria:

* Participants with a tinnitus diagnosis related to a Workman's Compensation Claim or any other litigation-related situation.
* Participants with tinnitus related to retrocochlear lesions, cochlear implants, or other unknown anatomic/structural lesions of the brain, skull base, temporal bone, or ear.
* Participants with hearing impairment such that they are unable to hear the highest volume of the computer cognitive training program.
* Participants with an active diagnosis of any acute or chronic central neurological condition including: Parkinson's disease, Multiple Sclerosis, Alzheimer's Disease, cerebral infarcts, traumatic brain injury, epilepsy, dementia, and/or a history of brain tumor(s).
* Subjects who have an active diagnosis of an anxiety disorder, psychosis or any psychiatric co-morbidity that may complicate the interpretation of study results.
* Participants with symptoms of severe depression on the Patient Health Questionnaire-9 (subjects who score >15 on the Patient Health Questionnaire-9 (PHQ-9) designed to screen for depression).
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year.
* Participants with kidney or liver impairment, a heart condition, porphyria, porphyria among family members, or an allergy to DCS.
* Participants who take any medication that is contraindicated with DCS.
* Use of any medications that may alter or affect cognition including, but not limited to, sedatives, hypnotics, narcotics, and opiates.
* Women who are pregnant or breast-feeding.
* People who have ever used the Brain Fitness Program® or any other computer based Brain Exercise or Brain Training programs within the prior year.
* Use of Neuromonics device for tinnitus treatment, or currently undergoing Tinnitus Retraining (TRT) program.
* Any condition the PI determines would render the study to not be in the best interest of the patient.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Tinnitus Handicap Inventory (THI) | Baseline and 5 weeks later
  We will measure THI before and after treatment. Primary efficacy is defined by a decrease of 17 points on their THI from baseline.

SECONDARY OUTCOMES:
Change in Neurocognitive assessment score | Baseline and 5 weeks later
  We will measure PASAT, Stroop, and a newly designed neurocognitive computer based test at the patient's baseline visit and final visit. These assessments are done as patients with tinnitus frequently report cognitive difficulties in attention and memory. One aim of this study is to target these cognitive difficulties. Improvements in memory and attention will be assessed using these neurocognitive tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Choi DC, Rothbaum BO, Gerardi M, Ressler KJ. Pharmacological enhancement of behavioral therapy: focus on posttraumatic stress disorder. Curr Top Behav Neurosci. 2010;2:279-99. doi: 10.1007/7854_2009_10. PMID 21309114
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Ganasen KA, Ipser JC, Stein DJ. Augmentation of cognitive behavioral therapy with pharmacotherapy. Psychiatr Clin North Am. 2010 Sep;33(3):687-99. doi: 10.1016/j.psc.2010.04.008. PMID 20599140
- [Background] Henry JA, Dennis KC, Schechter MA. General review of tinnitus: prevalence, mechanisms, effects, and management. J Speech Lang Hear Res. 2005 Oct;48(5):1204-35. doi: 10.1044/1092-4388(2005/084). PMID 16411806
- [Background] Kaltenbach JA. Neurophysiologic mechanisms of tinnitus. J Am Acad Audiol. 2000 Mar;11(3):125-37. PMID 10755809
- [Background] Lenarz T, Schreiner C, Snyder RL, Ernst A. Neural mechanisms of tinnitus. Eur Arch Otorhinolaryngol. 1993;249(8):441-6. doi: 10.1007/BF00168851. PMID 8442938
- [Background] Lockwood AH, Salvi RJ, Burkard RF. Tinnitus. N Engl J Med. 2002 Sep 19;347(12):904-10. doi: 10.1056/NEJMra013395. No abstract available. PMID 12239260
- [Background] Lockwood AH, Salvi RJ, Burkard RF, Galantowicz PJ, Coad ML, Wack DS. Neuroanatomy of tinnitus. Scand Audiol Suppl. 1999;51:47-52. PMID 10803913
- [Background] Shargorodsky J, Curhan GC, Farwell WR. Prevalence and characteristics of tinnitus among US adults. Am J Med. 2010 Aug;123(8):711-8. doi: 10.1016/j.amjmed.2010.02.015. PMID 20670725
- [Background] Siegmund A, Golfels F, Finck C, Halisch A, Rath D, Plag J, Strohle A. D-cycloserine does not improve but might slightly speed up the outcome of in-vivo exposure therapy in patients with severe agoraphobia and panic disorder in a randomized double blind clinical trial. J Psychiatr Res. 2011 Aug;45(8):1042-7. doi: 10.1016/j.jpsychires.2011.01.020. Epub 2011 Mar 5. PMID 21377691
- [Background] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Derived] Krings JG, Wineland A, Kallogjeri D, Rodebaugh TL, Nicklaus J, Lenze EJ, Piccirillo JF. A novel treatment for tinnitus and tinnitus-related cognitive difficulties using computer-based cognitive training and D-cycloserine. JAMA Otolaryngol Head Neck Surg. 2015 Jan;141(1):18-26. doi: 10.1001/jamaoto.2014.2669. PMID 25356570